CLINICAL TRIAL: NCT02393443
Title: The Effects of Oxytocin on Learning With Social Versus Nonsocial Motivation
Brief Title: Oxytocin and Learning for Teaching
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Matthew Lieberman, Matthew D. Lieberman, PhD, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 11-003565-1
Record Dates: First submitted 2015-01-22; First posted 2015-03-19 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Social Psychology
Keywords: oxytocin; healthy sample; intranasal administration; learning

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intranasal oxytocin (Experimental): Participants will self-administer 24 IU oxytocin (Syntocinon, Novartis Pharmaceuticals). 5 puffs per nostril (1 puff = 2.4 IU oxytocin).
  Interventions: Drug: Intranasal oxytocin
- Intranasal placebo (Placebo Comparator): 2 mls Glycerine and 3 mls purified water (methylparaben and propylparaben mixed according to purified water formula) for a total of 5 ml, which will be filtered with a 5mu filter. Participants will self-administer 5 puffs per nostril.
  Interventions: Drug: Intranasal placebo

INTERVENTIONS:
Drug: Intranasal oxytocin — Through the use of 1oz bottles attached with metered nasal pumps (1 puff = .1ml), participants will self-administer 24 IU oxytocin (Syntocinon, Novartis Pharmaceuticals). 5 puffs per nostril (1 puff = 2.4 IU oxytocin).
  Other Names: Syntocinon nasal spray
  Arms: Intranasal oxytocin
Drug: Intranasal placebo — Through the use of 1oz bottles attached with metered nasal pumps (1 puff = .1ml), participants will self-administer 5 puffs per nostril. Placebo consists of: 2 mls Glycerine and 3 mls purified water (methylparaben and propylparaben mixed according to purified water formula) for a total of 5 ml, which will be filtered with a 5mu filter.
  Arms: Intranasal placebo

SUMMARY:
One well-established cognitive theory propose a divide between social and non-social (i.e., cognitive) systems. However, recent work suggests that traditionally social systems can be utilized to enhance cognitive performance. In this study the investigators aim to explore this cooperation between oft-competing systems by instructing participants to learn information because they will be subsequently tested (the nonsocial learning-for-testing condition), or because they will be teaching the information to someone else (the prosocial learning-for-teaching condition). This latter condition relies upon the mentalizing system, which is used to contemplate another person's mental state, rather than traditional memory systems. This implies that the mnemonic powers of the mentalizing system can be leveraged in the learning of a broad array of non-social topics. Furthermore, there is also an emerging literature on the role of oxytocin, a neuropeptide naturally produced in the hypothalamus, in memory that parallels the social/nonsocial split. Oxytocin may benefit the learning-for-teaching group both in terms of enhancing initial social motivation and efficient use of the mentalizing system and then also in terms of memory consolidation for this information learning under socially-motivated conditions.

The investigators expect to replicate the basic learning-for-teaching effect such that those in the teaching condition will remember more than those in the testing conditions. They also expect an interaction between oxytocin administration and learning condition such that oxytocin administration should enhance learning for socially-motivated learning exclusively.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years of age
* Healthy (see below)
* Fluent in English
* Right-handed

Exclusion Criteria:

* Women who gave birth in the last six months, are currently pregnant, planning to become pregnant in the next 6 months, or currently breastfeeding women
* Symptoms of runny nose due to allergies/cold or other reason
* Current restricted fluid intake for any reason
* Heart disease
* Hypertension
* History of myocardial infarction
* History of cardiac arrhythmia
* Kidney or liver disease
* Vascular disease
* Epilepsy
* Migraine
* Asthma
* Nephritis
* Diabetes and other endocrine diseases
* Frequent or unexplained fainting
* History of stroke
* Aneurysm or brain hemorrhage
* Active psychiatric diagnosis
* Current psychopharmacologic treatment
* Drug or alcohol abuse
* Medical or neurological illness
* Regular use of medication (e.g., vasoconstrictive medications)
* Medication intake less than 2 weeks prior to study (5 weeks for fluoxetine) including daily non-steroidal anti-inflammatory drugs
* Smoking more than 15 cigarettes a day
* Consumption of any alcoholic beverages in the past 24 hours will be excluded
* Elevated blood pressure (>135/90)
* Low blood pressure (<90/55)
* Body temperature >100.1 F
* Left-handed
* Claustrophobia
* Presence of metal in their body

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 161 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Changes in brain neural activity, observed by fMRI, in response to a reading comprehension task | Between 40-90 minutes post administration
  Whole brain and region of interest (ROI) regression analysis will be used to compare the neural activity of participants in the tutor/memorizer and oxytocin/placebo groups. A design matrix will be created for each participant, modeling activity that is greater during reading comprehension compared with the grammar control passage. First level analyses will compare the response during the reading comprehension passages relative to the grammar control passages. Second level group analyses will compare the first level contrasts between the tutor vs. memorizer groups as well as the oxytocin vs. placebo groups. In regression analyses we will enter each participant's comprehension test score in the tutor and then memorizer condition as a regressor in a whole-brain and ROI analysis to determine which brain regions were more active during the encoding of the reading comprehension passage compared to the grammar control passage.

SECONDARY OUTCOMES:
Performance on a memory test of reading comprehension as measured by percentage of questions answered correctly | Between 40-90 minutes post administration
  Accuracy will be calculated for each participant by dividing the number of correct responses by the total number of questions. We will then conduct a between-subjects 2x2 ANOVA on the accuracy scores for the four groups of interest (i.e., oxytocin-tutor, oxytocin-memorizer, placebo-tutor, placebo-memorizer). A significance level of p<.05 will be used to determine whether there are significant differences between the groups. We will examine whether there is a main effect of either factor (oxytocin vs. placebo, tutor vs. memorize) as well as an interaction between the factors of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D Lieberman, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Department of Psychology, Los Angeles, California, United States

REFERENCES:
- [Derived] Straccia MA, Teed AR, Katzman PL, Tan KM, Parrish MH, Irwin MR, Eisenberger NI, Lieberman MD, Tabak BA. Null results of oxytocin and vasopressin administration on mentalizing in a large fMRI sample: evidence from a randomized controlled trial. Psychol Med. 2023 Apr;53(6):2285-2295. doi: 10.1017/S0033291721004104. Epub 2021 Oct 15. PMID 37310308